CLINICAL TRIAL: NCT05905991
Title: Feasibility and Efficacy of Enhanced Stress Resilience Training for Psychosocial and Occupational Wellbeing of Critical Care Nurses
Brief Title: Enhanced Stress Resilience Training for Critical Care Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CNR-2022-02
Record Dates: First submitted 2023-05-22; First posted 2023-06-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Job Stress; Burnout
Keywords: Burnout; Job stress; Resilience; Nurse; Critical care
MeSH Terms: conditions — Occupational Stress; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESRT Intervention (Experimental): Five 1-hour weekly ESRT sessions
  Interventions: Other: Enhanced Stress Resilience Training
- Waitlist Control (Other): The control group will receive ESRT after the intervention group finishes the 5-week ESRT program.
  Interventions: Other: Enhanced Stress Resilience Training

INTERVENTIONS:
Other: Enhanced Stress Resilience Training — The ESRT intervention will consist of 1) five weekly one-hour sessions (in-person or virtual) led by a certified instructor; 2) smartphone-based exercises that bring informal practice into daily life; 3) videos on principles and concepts taught each week; and 4) meditation recordings of various lengths and styles supporting the prescribed daily practice of up to 20 min/day. Weekly didactic and experiential activities will cover mindfulness-based intervention concepts and skills, such as cultivating resilience, awareness of the body, managing thoughts, responding versus reacting, transforming circumstances, and advocacy through mindful communication. The ESRT smartphone app ("Mindful Brian") houses all course materials (pre-class materials and post-class materials) and sends class reminders and messages. Considering nurses' shifts, ESRT will be offered in two separate sessions each week.

SUMMARY:
Job stress and burnout are significant problems affecting physical health, emotional well-being, job performance, and retention of nurses. Enhanced Stress Resilience Training (ESRT) is a theory-driven, evidence-based intervention to increase stress resilience and decrease burnout among clinicians. This study is a randomized waitlist-controlled trial to examine the efficacy, feasibility, and long-term sustainability of the 5-week ESRT intervention to improve psychosocial and occupational well-being of critical care nurses.

DETAILED DESCRIPTION:
The critical care setting is a stressful work environment where nurses provide intensive care to patients with life-threatening conditions. Regular job stress from the complex and fast-paced critical care work environment has been further intensified during the COVID-19 pandemic, which resulted in unprecedented challenges to health systems and has affected psychosocial and occupational wellbeing of healthcare workers. High or chronic job stress that is not properly managed can lead to burnout, which is characterized by emotional exhaustion, depersonalization, and decreased personal accomplishment. Burnout has negative impacts on physical and mental health (e.g., fatigue, anxiety, depression, sleep disorders), job performance or productivity (e.g., absenteeism, presenteeism), quality of care and patient care outcomes. Burnout also negatively affects nurses' retention and job turnover. The global prevalence of burnout among nurses ranges from 0.1% to 47.8% (pooled prevalence 11.2%) and critical care nurses are reported to have the highest prevalence of burnout (14.4%) among all specialties. Therefore, there is a substantial need to address burnout and promote occupational wellness of critical care nurses. Enhanced Stress Resilience Training (ESRT) is a theory-driven, evidence-based intervention developed by UCSF Associate Professor of Surgery, Dr. Carter Lebares aimed at increasing stress resilience and decreasing burnout among clinicians. The purpose of this study is to examine the efficacy, feasibility, and long-term sustainability of the 5-week ESRT intervention to improve psychosocial and occupational well-being among critical care nurses. The study will conduct a randomized waitlist-controlled trial among 100 UCSF critical care nurses.

ELIGIBILITY:
Inclusion Criteria:

* Adult critical care nurses employed at UCSF Health.

Exclusion Criteria:

* Those who cannot commit to participation in all five ESRT sessions
* Temporary travel nurses.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in burnout score | Baseline to immediately post-ESRT intervention; Baseline to 1 month after ESRT intervention; Baseline to 3 months after ESRT intervention
  A 9-item short version of the Maslach Burnout Inventory-Human Services Survey (MBI-HSS) will be used. The MBI-HSS has 3 subscales of emotional exhaustion (EE, 3 items), depersonalization (DP, 3 items), and personal accomplishment (PA, 3 items). Each subscale is measured by 7-point response categories (1=Never ~ 4= A few times a month ~ 7=Every day). Higher scores of EE and DP and a lower score of PA indicated higher burnout.

SECONDARY OUTCOMES:
Changes in mindfulness score | Baseline to immediately post-ESRT intervention; Baseline to 1 month after ESRT intervention; Baseline to 3 months after ESRT intervention
  Mindfulness reflects the mental skills of attention, emotional regulation and metacognition and will be measured by the 10-item Cognitive Affective Mindfulness Scale-Revised (CAMS-R). Response categories include 1=rarely/not at all, 2=sometimes, 3=often, 4=almost always. Higher scores indicate higher mindfulness.
Changes in resilience score | Baseline to immediately post-ESRT intervention; Baseline to 1 month after ESRT intervention; Baseline to 3 months after ESRT intervention
  Resilience refers to "an ability to bounce back or recover from stress" and will be measured by the 6-item Brief Resilience Scale (BRS). 5-point Likert response categories are used: 1=Strongly disagree to 5=Strongly agree. Three items are negatively worded, and the scores of these items will be reverse-coded. Higher scores indicate higher resilience.
Changes in work ability score | Baseline to immediately post-ESRT intervention; Baseline to 1 month after ESRT intervention; Baseline to 3 months after ESRT intervention
  Physical and mental work ability will be assessed by three questions from the Work Ability Scale: (1) Current work ability compared to your highest work ability ever (0=cannot work at all ~ 10=able to work at my best), (2) current ability to work with respect to the physical job demands (poor, fair, good, very good, excellent), (3) current ability to work with respect to the mental job demands (poor, fair, good, very good, excellent). Higher scores indicate higher work ability.
Changes in professional fulfillment index score | Baseline to immediately post-ESRT intervention; Baseline to 1 month after ESRT intervention; Baseline to 3 months after ESRT intervention
  Professional Fulfillment Index (PFI) will be measured by the 6-item Professional Fulfillment Subscale (0=not at all true to 4=completely true). The PFI score is calculated by averaging the item scores and ranges from 0 to 4. Higher scores indicate higher professional fulfillment.
Changes in psychological safety score | Baseline to immediately post-ESRT intervention; Baseline to 1 month after ESRT intervention; Baseline to 3 months after ESRT intervention
  The Psychological Safety Scale (10 items) will be used to measure psychological safety. The response format uses a 5-point Likert scale (1=Strongly disagree to 5=Strongly agree). Higher scores indicate higher psychological safety.
Percentage of participants who are satisfied with the job | Baseline, immediately post-ESRT intervention, 1-month and 3-month after ESRT intervention
  Job satisfaction will be asked by one question: How satisfied are you with your current job in this hospital? The 4-point Likert-Type response format (Very dissatisfied, A little dissatisfied, Moderately satisfied, Very satisfied) will be used. The response will be dichotomized into dissatisfied and satisfied.
Changes in perceived stress score | Baseline to immediately post-ESRT intervention; Baseline to 1 month after ESRT intervention; Baseline to 3 months after ESRT intervention 3-month after the 5-week ESRT
  Perceived stress will be measured by Cohen's Perceived Stress Scale (PSS), which includes 10 items and uses a 5-point response format (1=never to 5=very often). Higher scores indicate higher stress.
Changes in depressive symptom score | Baseline to immediately post-ESRT intervention; Baseline to 1 month after ESRT intervention; Baseline to 3 months after ESRT intervention th, and 3-month after the 5-week ESRT
  Depressive symptoms will be measured by the Patient Health Questionnaire-8 (PHQ-8) using 4-point response format (1=not at all to 4=nearly every day). Higher scores indicate higher depression.
Percentage of participants who have the intention to leave the job | Baseline, immediately post-ESRT intervention, 1-month and 3-month after ESRT intervention
  Intention to leave the job will be measure by the question "How likely are your to leave your current position in the next year?" using a 7-point Likert-Type response format (7=Definitely leaving ~ 4=Neutral ~ 1=Not leaving). Responses will be dichotomized: 1-4 Not leaving and 5-7 Having the intention to leave the job

OTHER OUTCOMES:
Percentage of participants in each ESRT session | 5-week intervention period
  The number of participants in each weekly session and the number of sessions that each subject attends will be observed and recorded.
ESRT acceptability scores | Immediately post-ESRT intervention, 1-month and 3-month after ESRT intervention
  ESRT acceptability will be measured by the 6-item Credibility-Expectancy Questionnaire (CEQ) and one question "I would recommend this course to a peer". Response formats are 0-10 or 0-100%. Higher scores indicate higher acceptability.
The frequency of ESRT skill use (ESRT sustainability) | Immediately post-ESRT intervention, 1-month and 3-month after ESRT intervention
  Participants will be asked about the frequency of ESRT skill use (daily, several times a week, several times a month, rarely, never). The frequency will be described by the count and percentage by category.

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Jeong Lee, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghawadra SF, Abdullah KL, Choo WY, Phang CK. Mindfulness-based stress reduction for psychological distress among nurses: A systematic review. J Clin Nurs. 2019 Nov;28(21-22):3747-3758. doi: 10.1111/jocn.14987. Epub 2019 Jul 22. PMID 31267619
- [Background] Kleinpell R, Moss M, Good VS, Gozal D, Sessler CN. The Critical Nature of Addressing Burnout Prevention: Results From the Critical Care Societies Collaborative's National Summit and Survey on Prevention and Management of Burnout in the ICU. Crit Care Med. 2020 Feb;48(2):249-253. doi: 10.1097/CCM.0000000000003964. PMID 31939795
- [Background] Lebares CC, Guvva EV, Olaru M, Sugrue LP, Staffaroni AM, Delucchi KL, Kramer JH, Ascher NL, Harris HW. Efficacy of Mindfulness-Based Cognitive Training in Surgery: Additional Analysis of the Mindful Surgeon Pilot Randomized Clinical Trial. JAMA Netw Open. 2019 May 3;2(5):e194108. doi: 10.1001/jamanetworkopen.2019.4108. PMID 31125095
- [Background] Lebares CC, Hershberger AO, Guvva EV, Desai A, Mitchell J, Shen W, Reilly LM, Delucchi KL, O'Sullivan PS, Ascher NL, Harris HW. Feasibility of Formal Mindfulness-Based Stress-Resilience Training Among Surgery Interns: A Randomized Clinical Trial. JAMA Surg. 2018 Oct 1;153(10):e182734. doi: 10.1001/jamasurg.2018.2734. Epub 2018 Oct 17. PMID 30167655
- [Background] Shah MK, Gandrakota N, Cimiotti JP, Ghose N, Moore M, Ali MK. Prevalence of and Factors Associated With Nurse Burnout in the US. JAMA Netw Open. 2021 Feb 1;4(2):e2036469. doi: 10.1001/jamanetworkopen.2020.36469. PMID 33538823
- [Background] Lebares CC, Guvva EV, Desai A, Herschberger A, Ascher NL, Harris HW, O'Sullivan P. Key factors for implementing mindfulness-based burnout interventions in surgery. Am J Surg. 2020 Feb;219(2):328-334. doi: 10.1016/j.amjsurg.2019.10.025. Epub 2019 Oct 17. PMID 31668282
- [Background] Sulosaari V, Unal E, Cinar FI. The effectiveness of mindfulness-based interventions on the psychological well-being of nurses: A systematic review. Appl Nurs Res. 2022 Apr;64:151565. doi: 10.1016/j.apnr.2022.151565. Epub 2022 Jan 15. PMID 35307128
- [Background] Woo T, Ho R, Tang A, Tam W. Global prevalence of burnout symptoms among nurses: A systematic review and meta-analysis. J Psychiatr Res. 2020 Apr;123:9-20. doi: 10.1016/j.jpsychires.2019.12.015. Epub 2020 Jan 22. PMID 32007680